CLINICAL TRIAL: NCT06442696
Title: Effect Of Healthy Choices Program On Nutrition, Physical Activity And Body Mass Index In Adolescents
Brief Title: Effect Of HCP On Nutrition, Physical Activity And Body Mass Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tugba Duygu Ozmet, Instructor, Bahçeşehir University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 123
Record Dates: First submitted 2024-02-07; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Obesity; Adolescent Obesity
Keywords: School nursing; Healthy choices; Nutrition; Physical Activity
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 10-14 years old adolescent are given health education Health education was given
  Interventions: Other: Health Education: Healthy Choices Program
- Control Group (No Intervention): 10-14 years old adolescent are not given health education

INTERVENTIONS:
Other: Health Education: Healthy Choices Program — Six session for students and school personel
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to test effectiveness of "The Healthy Choices Program, in adolescents. The main question[s] it aims to answer are:

1. Effectiveness of Healthy Choices on Body Mass Index
2. Effectiveness of Healthy Choices on Health Attitude, Nutrition and Physical Activity Knowledge
3. Effectiveness of Healthy Choices on Fruit,vegetable, water consumption

DETAILED DESCRIPTION:
In our study, a quasi-experimental design with a pre-test and post-test control group was used. This study was carried out between May 2022 and January 2023. 150 adolescents in the 5th, 6th and 7th grades of two secondary schools in Istanbul were included in the study. One of the schools was designated as the intervention group (n=75) and the other as the control group (n=75). Six sessions of training were given to the intervention group. Data were collected using the Descriptive Characteristics Form, Healthy Habits Questionnaire, Adolescent Attitude Scale, Adolescent Physical Activity Knowledge Scale, Adolescent Nutrition Knowledge Scale and Physical Activity Questionnaire. Chi-square test, t test, Mann-Whitney U test, Wilcoxon test were used to analyze the data.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents in 6th, 7th and 8th grades

  * Adolescents without mental disabilities
  * Families and adolescents who agree to participate in the study

Exclusion Criteria:

* Families and adolescents who did not agree to participate in the study were not included in the study.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Increasing consumption of fruit and vegetables in the experimental group | Up to six months
  It was measured by using Healthy Habits Questionnaire. (Item 1:How many servings of ruits or vegetables do you eat a day? (One serving is most easily identified by the size of the palm of your hand.) There is no scoring for this questionnaire.
Decreasing screen time of adolescents in the experimental group | Up to six months
  It was measured by using the Healthy Habits Questionnaire. (Item 5:How many hours a day do you watch TV/movies or sit and play video/computer games? There is no scoring for this questionnaire.)
Increasing physical activity level of adolescents in the experimental group | Up to six months
  It was measured using the Healthy Habits and Physical Activity Questionnaire. In Healthy Habits Questionnaire Item 8:How much time a day do you spend in active play (faster breathing/heart rate or sweating)? was used. The Physical Activity Questionnaire is a 7-day recall-based measurement tool designed to assess overall physical activity levels throughout the school year.The minimum score for each item of the questionnaire is 1 and the maximum score is 5. The minimum score to be obtained from questionnaire is 9 and the maximum score is 45. Item 10 is not included in scoring.
Decreasing consumption sugary drinks of adolescents in the experimental group | Up to six months
  It was measured by Healthy Habits Questionnaire (Item 9:How How many 8-ounce servings of the following do you drink a day (soda,fruit juice,sport drinks)

SECONDARY OUTCOMES:
Increasing consumption water and milk of adolescents in the experimental group | Up to six months
  It was measured by using Healthy Habits Questionnaire (Item 9:How many 8-ounce servings of the following do you drink water/milk a day?)There is no scoring for this questionnaire.
Increasing healthy lifestyle attitude scale score of adolescents in the experimental group | Up to six months
  It was measured using the healthy lifestyle attitude scale. The scale was composed of 14 items to determine adolescents' attitudes toward nutrition, physical activity, and sleep behavior. The responses are scored on a 5-point Likert-type scale ranging from strongly disagree (1) to agree (5) strongly. The Cronbach's alpha of the original scale is 0.84 and the item-total score correlations are between 0.43 and 0.68 .
Increasing adolescent nutrition knowledge of adolescents in the experimental group | Up to six months
  It was measured using the adolescent nutrition knowledge scale. The scale consisted of 20 items and was developed to determine the level of knowledge about nutrition in adolescents, such as the types of nutrients, portion size, and eating habits. The answer categories of each question are structured as "yes", "no" or "do not know". The Cronbach's alpha of the original scale is 0.86, and item-total score correlations are between 0.13 and 0.59.
Increasing Adolescent activity knowledge of adolescents in the experimental group | Up to six months
  It was measured using the adolescent activity knowledge scale. The Activity Scale consists of 12 items and was developed to determine the knowledge level of physical activity and exercise in adolescents. The answers categories of each question are structured as "yes", "no", and "do not know". The Cronbach's alpha of the original scale is 0.69, and item-total score correlations are between 0.22 and 0.46.
Reducing Body Mass Index of adolescents in the experimental group | Up to six months
  The weight and height of adolescents were measured by the researcher. Tanita Bc-730 was used as a weighing machine. Mesilife Mst-200 was used as a height meter. They were measured in schools. After, body mass indexes were calculated for each adolescent.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba D Ozmet, PhD, Principal Investigator — Bahçeşehir University; Tugba D Ozmet, PhD, Study Chair — Bahçeşehir University
Locations (1):
- Tugba Duygu OZMET, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No